CLINICAL TRIAL: NCT04100889
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Alzheimer's Disease
Status: Withdrawn | Type: Observational
Why Stopped: Company focus shifted
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-007
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2021-09

CONDITIONS: Alzheimer Disease; Alzheimer Disease 1; Alzheimer Disease 2; Alzheimer Disease 3; Alzheimer Disease 4; Alzheimer Disease 5; Alzheimer Disease 6; Alzheimer Disease 7; Alzheimer Disease 8; Alzheimer Disease 9, Late-Onset; Alzheimer Disease 10; Alzheimer Disease 11; Alzheimer Disease 12; Alzheimer Disease 13; Alzheimer Disease 14; Alzheimer Disease 15; Alzheimer Disease 16; Alzheimer Disease 17; Alzheimer Disease 18; Alzheimer Disease 19; Alzheimer Disease, Early Onset; Alzheimer Disease, Late Onset; Alzheimer Disease Focal
Keywords: Microbiome
MeSH Terms: conditions — Alzheimer Disease; Alzheimer disease type 1; Alzheimer disease type 2; Alzheimer disease, familial, type 3; Alzheimer disease type 4; Alzheimer Disease 5; Alzheimer Disease 6; Alzheimer Disease 7; Alzheimer Disease 8; Alzheimer Disease 9; Alzheimer Disease 10; Alzheimer Disease 11; Alzheimer Disease 12; Alzheimer Disease 13; Alzheimer Disease 14; Alzheimer Disease 15; Alzheimer Disease 16

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Alzheimer's disease patients: Patients who have been diagnosed with Alzheimer's disease
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention for this study.

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records regarding Alzheimer's disease.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records regarding Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
2. Male or female patients age 18 and older
3. Diagnosis of Alzheimer's disease or dementia by a physician
4. Mini Mental Status Exam score less than 26

Exclusion Criteria:

1. Refusal to sign informed consent form
2. Treatment with antibiotics within 2 weeks prior to screening
3. Treatment with probiotics within 2 weeks prior to screening
4. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
5. Postoperative stoma, ostomy, or ileoanal pouch
6. Participation in any experimental drug protocol within the past 12 weeks
7. Treatment with total parenteral nutrition
8. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
9. Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age or older and have been diagnosed with Alzheimer's disease.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Alzheimer's Disease via Relative Abundance Found in Microbiome Sequencing | 1 year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be correlated to Alzheimer's disease state

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only aggregated and deidentified data will be shared with other researchers